CLINICAL TRIAL: NCT00572728
Title: 3'-Deoxy-3'-18F Fluorothymidine PET/CT in Predicting Response To Chemotherapy Before Surgery in Patients With Locally Advanced Breast Cancer
Brief Title: Phase II Study of Fluorine-18 3'-Deoxy-3'-Fluorothymidine (F-18-FLT) in Invasive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2009-00266; NCI-2009-00266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACRIN 6688 (Other: American College of Radiology Imaging Network); 8029 (Other: CTEP); N01CM27165 (NIH); NCT00566293 (obsolete NCT alias)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (18F-FLT) (Experimental): Patients undergo 18F-FLT PET /CT at baseline (prior to chemotherapy, FLT-1), early therapy (5-10 days after the initiation of the first course of chemotherapy, FLT-2), and post therapy (within 3 weeks prior to surgery, FLT-3). Patients undergo standard surgical resection of residual tumor following completion of neoadjuvant chemotherapy.
  Interventions: Procedure: CT; Drug: 18F-FLT; Procedure: PET

INTERVENTIONS:
Procedure: CT — Undergo 18F-FLT PET/CT
  Other Names: CAT; CAT Scan; Computed Tomography; Computerized Axial Tomography; Computerized Tomography; CT SCAN; tomography
Drug: 18F-FLT — Undergo 18F-FLT PET/CT
  Other Names: Fluorothymidine F-18; 3'-deoxy-3'-(18F) fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F 18
Procedure: PET — Undergo 18F-FLT PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; Positron Emission Tomography; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well 3'-deoxy-3'-18F fluorothymidine (18F-FLT) positron emission tomography (PET)/computed tomography (CT) works in predicting response in patients receiving chemotherapy and undergoing surgery for breast cancer that has spread from where it started to nearby tissue or lymph nodes. Diagnostic procedures, such as 18F-FLT PET/CT, may help in learning how well chemotherapy works to kill breast cancer cells before surgery and help doctors plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To correlate the percentage change in standardized uptake value at 60 minutes (SUV60) between baseline (FLT-1) and early-therapy (FLT-2) with pathologic complete response to neoadjuvant chemotherapy of the primary tumor in patients with locally advanced breast cancer.

SECONDARY OBJECTIVES:

I. To demonstrate correlation between FLT-1 and post-therapy (FLT-3) uptake parameters and tumor proliferation markers in locally advanced breast cancer.

II. To evaluate the relationship between FLT-1, FLT-2 and FLT-3 uptake parameters and pathologic complete response of the primary tumor and residual cancer burden (RCB).

III. To evaluate the relationship between FLT-1, FLT-2 and FLT-3 uptake parameters and non-response of the primary tumor (stable or progressive disease) to therapy.

IV. To evaluate the relationship between FLT-1, FLT-2 and FLT-3 uptake parameters and pathologic complete response to neoadjuvant chemotherapy in patients with regional disease in the lymph nodes in patients with locally advanced breast cancer.

V. To compare the changes of FLT-2 and FLT-3 uptake parameters to changes in tumor sizes from other serial imaging modalities such as mammograms, magnetic resonance imaging (MRI), and ultrasound.

VI. To compare the changes of FLT-2 and FLT-3 uptake parameters to metabolic changes from [18F] fludeoxyglucose (FDG)-PET, as available.

VII. To continue to monitor for potential safety issues and define any physiologic effects associated with 18F FLT administration.

OUTLINE:

Patients undergo 18F-FLT PET/CT at baseline (prior to chemotherapy, FLT-1), early therapy (5-10 days after the initiation of the first course of chemotherapy, FLT-2), and post therapy (within 3 weeks prior to surgery, FLT-3). Patients undergo standard surgical resection of residual tumor following completion of neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed breast cancer, determined to be a candidate for primary systemic (neoadjuvant) therapy and for surgical resection of residual primary tumor following completion of neoadjuvant therapy
* Locally advanced breast cancer, not stage IV, and with a tumor size >= 2 cm (as measured on imaging or estimated by physical exam)
* No obvious contraindications for primary chemotherapy
* Residual tumor planned to be removed surgically following completion of neoadjuvant therapy
* Able to lie still for 1.5 hours for PET scanning
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times the institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* If female, postmenopausal for a minimum of one year, OR surgically sterile, OR not pregnant, confirmed by institutional standard of care (SOC) pregnancy test, and willing to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation
* Able to understand and willing to sign a written informed consent document and a Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines

Exclusion Criteria:

* Previous treatment (chemotherapy, radiation, or surgery) to involved breast; including hormone therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Medically unstable
* Condition requiring anesthesia for PET scanning and/or unable to lie still for 1.5 hours
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to F-18 fluorothymidine
* Pregnant or nursing
* Previous malignancy, other than basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix, from which the patient has been disease free for less than 5 years
* Currently on hormone therapy as the primary systemic neoadjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lale Kostakoglu, Principal Investigator — American College of Radiology Imaging Network
Locations (27):
- United States (27):
  - Scottsdale Medical Imaging Limited, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Morton Plant Hospital, Clearwater, Florida
  - Morton Plant Mease, Dunedin, Florida
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Radiology Consultants Inc, Youngstown, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - American College of Radiology Imaging Network, Philadelphia, Pennsylvania
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Excel Diagnostics, Houston, Texas
  - Westchase Oncology Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Result] Kostakoglu L, Duan F, Idowu MO, Jolles PR, Bear HD, Muzi M, Cormack J, Muzi JP, Pryma DA, Specht JM, Hovanessian-Larsen L, Miliziano J, Mallett S, Shields AF, Mankoff DA; ACRIN 668 Investigative Team. A Phase II Study of 3'-Deoxy-3'-18F-Fluorothymidine PET in the Assessment of Early Response of Breast Cancer to Neoadjuvant Chemotherapy: Results from ACRIN 6688. J Nucl Med. 2015 Nov;56(11):1681-9. doi: 10.2967/jnumed.115.160663. Epub 2015 Sep 10. PMID 26359256
- See also: A Phase II Study of [(18)F]-3'Deoxy-3'-Fluorothymidine Positron Emission Tomography (FLT-PET) in The Assessment of Early Response of Breast Cancer to Neoadjuvant Chemotherapy: Results From ACRIN 6688 — http://jnm.snmjournals.org/content/early/2015/09/09/jnumed.115.160663.long

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (18F-FLT): Patients undergo 18F-FLT PET/CT at baseline (prior to chemotherapy, FLT-1), early therapy (5-10 days after the initiation of the first course of chemotherapy, FLT-2), and post therapy (within 3 weeks prior to surgery, FLT-3). Patients undergo standard surgical resection of residual tumor following completion of neoadjuvant chemotherapy.
  Fluorothymidine F-18: Undergo 18F-FLT PET/CT
  Positron Emission Tomography: Undergo 18F-FLT PET/CT
  Computed Tomography: Undergo 18F-FLT PET/CT
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Diagnostic (18F-FLT)
Started | 90 (Registered)
Eligible | 87
Enrolled Under Amendment 5 or Later | 82
Did Not Withdraw | 72
On Study | 71
Completed FLT1 Scan | 67
First Therapy Initiated | 65
Completed FLT2 Scan | 60
Second Chemotherapy Initiated | 59
Second Chemotherapy Initiated After FLT2 | 52
Pathology Complete | 51
Completed FLT3 Scan | 43 (Secondary analysis milestone: 43 pts had FLT-3 performed.)
LN Evaluation After NAC | 38 (Secondary:38 patients were available for histopathological LN evaluation after NAC)
RCB Evaluation | 35 (Secondary: histopathology was available in 35 patients for RCB evaluation)
Completed | 51 (51 patients eligible for primary objective analysis)
Not Completed | 39
Not completed — Withdrawal by Subject | 10
Not completed — Ineligible | 3
Not completed — Enrolled under Amendment 4 | 5
Not completed — Offstudy due to complicating disease | 1
Not completed — FLT1 not completed | 4
Not completed — First Chemotherapy not initiated | 2
Not completed — FLT2 not completed | 5
Not completed — Second chemotherapy not initiated | 1
Not completed — FLT2 after second chemotherapy initiated | 7
Not completed — Pathology missing | 1

BASELINE CHARACTERISTICS:
Population: Registered
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 90
Age, Continuous [Mean (Full Range); unit: years] | 51 [22 to 83]
Gender [Count of Participants; unit: Participants] — Overall Number of Baseline Participants
  Participants
    Female | 90
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 51
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: %Change in FLT Uptake Between the Baseline (Pre-therapy) and the Early-therapy Imaging Studies to Predict Pathological Complete Response
Description: The primary statistical evaluation will be based on the percent change in FLT SUV60 between baseline (pre-therapy, FLT-1) and the early-therapy imaging (5-10 days after chemotherapy, FLT-2) studies
Time Frame: Baseline (FLT-1) to early therapy (5-10 days after chemotherapy, FLT-2)
Population: Percent Change in Maximum Standardized FLT uptake between the baseline (pre-therapy, FTL-1) and the early-therapy imaging (5-10 days after chemotherapy, FLT-2)
Measure: Mean (Standard Deviation); unit: percentage change of SUVmax
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 51
percentage change of SUVmax | 38.78 (26.07)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); A receiver operating characteristic (ROC) analysis was performed to assess the significance of the Area Under the Curve (AUC) under the Null Hypothesis with a one sided alpha=0.05 (95% one-sided CL): H0: AUC = 0.50 (no difference from guessing) given the alternative hypothesis: Ha:AUC >= 0.75 AUC = ROC(%ΔSUVmax| path response) where percent change (%ΔSUVmax ) was defined as (SUVmax at FLT1 -SUVmax at FLT2)/SUVmax at FLT1 x 100; Test type: Superiority or Other; p = 0.046, Delong method — The Delong method was used to test if the observed AUC was significantly different than 0.5 with the one-sided p value DeLong ER, DeLong DM, Clarke-Pearson DL, Biometrics (1988); one-sided p-value; AUC = 0.68, 95% CI 1-sided [upper limit .83], Standard Error of Mean 0.10 — percent change in SUVmax was computed as: %ΔSUVmax = 100*(FLT1-FLT2)/FLT1 a 90% 2-sided confidence interval was constructed from 2000 Bootstrapping estimates from which the 1-sided 95% CI was derived. Hanley SE(AUC) reported

2. Secondary Outcome: Correlation Between SUVmax and Ki-67 LI at FLT1(Baseline PET)
Description: For the purposes of reporting, SUVmax @ FLT1 will be considered the outcome. the correlation is measured between the fraction of Ki-67-positive tumor cells (the Ki-67 labeling index) and SUVmax at FLT1 .
  Ki-67 labeling index (LI) was calculated as the number of Ki-67 positive tumor cells per one thousand tumor cells.
Time Frame: Baseline (FLT-1)
Population: 1 of the 73 participants did not have both FLT-1 and Ki-67 LI available data
Measure: Mean (Standard Deviation); unit: Standard Uptake Values (SUVmax)
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 72
Standard Uptake Values (SUVmax) | 5.71 (3.20)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); H0: ρ = 0; that is, there is no correlation between SUVmax @ FLT-1 and Ki-67 LI a Fisher's z Transformation was applied to adjust for bias in the Spearman Correlation Statistic; Test type: Superiority or Other; p = 0.002, spearman correlation method; spearman correlation = 0.35, 95% CI 2-sided [0.13 to 0.54] — This estimate uses the Fisher's z Transformation to adjust for bias in the Spearman Correlation Statistic

3. Secondary Outcome: Correlation Between SUVmax and Ki-67 LI at FLT3 (Post-NAC)
Description: For the purposes of reporting, SUVmax @ FLT-3 will be considered the outcome. correlation between the fraction of Ki-67-positive tumor cells (the Ki-67 labeling index) and SUVmax at FLT-3 Ki-67 labeling index (LI) was calculated as the number of Ki-67 positive tumor cells per one thousand tumor cells.
Time Frame: Post-NAC (FLT3)
Population: 43 patients who had suitable post-NAC tissue samples for correlation between surgical specimens and FLT3 SUVs
Measure: Mean (Standard Deviation); unit: Standard Uptake Values (SUVmax)
Groups:
- Diagnostic (18F-FLT): Patients undergo 18F-FLT PET/CT at baseline (prior to chemotherapy, FLT-1), early therapy (5-10 days after the initiation of the first course of chemotherapy, FLT-2), and post-NAC (within 3 weeks prior to surgery, FLT-3). Patients undergo standard surgical resection of residual tumor following completion of neoadjuvant chemotherapy.
  Fluorothymidine F-18: Undergo 18F-FLT PET/CT
  Positron Emission Tomography: Undergo 18F-FLT PET/CT
  Computed Tomography: Undergo 18F-FLT PET/CT
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 43
Standard Uptake Values (SUVmax) | 1.88 (1.88)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); H0: ρ = 0; that is, there is no correlation between SUVmax @ FLT-3 and Ki-67 LI; Test type: Superiority or Other; p < 0.0001, Spearman Correlation method; we use Fisher's z Transformation to adjust for bias in the Spearman Correlation Statistic; Spearman Correlation = 0.67, 95% CI 2-sided [0.47 to 0.81] — this estimate uses the Fisher's z Transformation to adjust for bias in the Spearman Correlation Statistic

4. Secondary Outcome: SUVmax at FLT-1 Comparison Between Residual Cancer Burden (RCB) 0/I and RCB II/III
Description: While normally RCB (or other final determination) would be considered the outcome, since this is a predictive question, we will consider the Standardized Uptake Values the measurement of interest and report those values herein.
  Mean Standard Uptake Values (max) at Baseline (FLT-1) were compared for Participants with Residual Cancer Burden 0/I vs Residual Cancer Burden of II/III
Time Frame: Baseline (FLT-1)
Population: @ Baseline: 35 patients with FLT-1 were evaluable for RCB: 14 patients with RCB 0/I and 21 patients with RCB II/III
Measure: Mean (Standard Deviation); unit: Standard Uptake Values (SUVmax)
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 35
Standard Uptake Values (SUVmax)
  All Data | 5.9 (3.2)
  RCB 0,I | 6.2 (2.9)
  RCB II,III | 5.8 (3.5)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); H0: Mean SUVmax (RCB 0,I) = Mean SUVmax (RCB II,III) After dichotomization, Wilcoxon two-sample test was used to compare uptake values between RCB groups. In other words, we are comparing the means (of SUVmax) @ FLT1 between the RCB 0,I and the RCB II,III groups; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney); two-sided exact p value from Wilcoxon two-sample test

5. Secondary Outcome: SUVmax at FLT-2 Comparison Between Residual Cancer Burden (RCB) 0/I and RCB II/III
Description: While normally RCB (or other final determination) would be considered the outcome, since this is a predictive question, we will consider the uptake values the measurement of interest and report those values herein.
  Mean Standard Uptake Values (max) after one cycle of NAC (FLT2) were compared for Participants with Residual Cancer Burden (RCB) 0/I vs RCB II/III
Time Frame: early treatment (FLT2)
Population: after one cycle of NAC (FLT2): 35 patients had FLT-2 and RCB evaluation: 14 patients with RCB 0/I and 21 patients with RCB II/III
Measure: Mean (Standard Deviation); unit: Standard Uptake Values (SUVmax)
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 35
Standard Uptake Values (SUVmax)
  All Data | 3.3 (2.0)
  RCB 0,I | 3.5 (2.3)
  RCB II,III | 3.2 (1.9)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); H0: SUVmax (RCB 0,I) = SUVmax (RCB II,III) in other words, we are comparing the SUVmax @ FLT2 between the RCB 0,I and the RCB II,III groups; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney); *two-sided exact p value from Wilcoxon two-sample test

6. Secondary Outcome: SUVmax at FLT-3 Comparison Between Residual Cancer Burden (RCB) 0/I and RCB II/III
Description: The Standard Uptake Values (max) after completion of NAC (FLT-3) were compared for Participants with Residual Cancer Burden 0/I vs Residual Cancer Burden of II/III While normally RCB (or other final determination) would be considered the outcome, since this is a predictive question, we will consider the mean of the uptake values the measurement of interest and report those values herein.
Time Frame: post-NAC (FLT-3)
Population: After completion of NAC (FLT-3): only 31 patients had both FLT3 and RCB evaluation: 11 patients with RCB 0/I and 20 patients with RCB II/III
Measure: Mean (Standard Deviation); unit: Standard Uptake Values (SUVmax)
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 31
Standard Uptake Values (SUVmax)
  All Data (FLT3) | 1.8 (1.8)
  RCB 0/I (FLT3) | 0.7 (0.3)
  RCB II/III (FLT3) | 2.4 (2.0)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); H0: SUVmax (RCB 0,I) = SUVmax (RCB II,III) in other words, we are comparing the SUVmax @ FLT3 between the RCB 0,I and the RCB II,III groups; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney); two-sided exact p value from Wilcoxon two-sample test
Statistical Analysis 2: Comparison: Diagnostic (18F-FLT); H0: %SUVmax FLT1-FLT3 (RCB 0,I) = %SUVmax FLT1-FLT3 (RCB II,III) A logistic regression model is used to determine if a larger percent change in SUVmax is associated with (RCB 0,I); the null hypothesis assumes that there is no association; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.76 to 0.97]

7. Secondary Outcome: Change in Uptake Between FLT1 and FLT3 to Predict Pathologic Complete Response (pCR) of the Primary Tumor
Description: To evaluate the relationship between the change in uptake between FLT1 and FLT3 and pathologic complete response, an ROC curve will be estimated and the area under the curve (AUC), along with its 90% confidence interval, will be determined. For the purposes of reporting, we will consider the percent change in uptake between FLT1 and FLT3 to be the outcome.
  Reported values in the Outcome Measure table represent Change in uptake between FLT1 and FLT3, i.e., percentage change of SUVmax. The relationship between the change in uptake between FLT1 and FLT3 and pathological complete response was assessed by using ROC analysis. The Area Under the ROC Curve is reported in the Statistical Analysis section
Time Frame: Baseline (FLT-1) and post-NAC (FLT-3)
Population: 43 patients who had both FLT1 and FLT3 scans
Measure: Mean (Standard Deviation); unit: percentage change in SUVmax
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 43
percentage change in SUVmax
  All Data | 38.8 (26.1)
  pCR | 52.7 (22.8)
  no-pCR | 35.8 (26.0)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); ROC analysis was used to compute the AUC and evaluate if %ΔSUVmax FLT1-FLT3 is predictive of pCR with alpha=0.05. The Null Hypothesis assumes that the P(%ΔSUVmax FLT1-FLT3|pCR)= 1 - P(%ΔSUVmax FLT1-FLT3|non-pCR) that is: H0: AUC =0.5 (guessing); Test type: Superiority or Other; p < 0.001, Delong Method — Delong 1-sided p-value (alpha=0.05); The Delong-Delong Clark-Pearson method using modified U-statistics was used to evaluate the AUC; AUC = 0.83, 90% CI 2-sided [.72 to .94]

8. Secondary Outcome: %Change SUVmax From FLT1-FLT2 to Predict Lymph Node Status at Surgery
Description: Reported values in the Outcome Measure table represent %Change in uptake between FLT1 and FLT2, i.e., percentage change of SUVmax. The relationship between the change in uptake between FLT1 and FLT2 and lymph node (LN) status. For the purposes of reporting, the % Change in SUV will be considered the outcome.
Time Frame: Baseline (FLT-1) and Early Therapy (FLT-2)
Population: Data on 38 patients having FLT1 and FLT2 were available for histopathological LN evaluation after NAC: 14 with negative nodes, 15 with 1-3 LN metastases and 9 with >3 LN metastases
Measure: Mean (Standard Deviation); unit: percent change in SUVmax from FLT1-FLT2
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 38
percent change in SUVmax from FLT1-FLT2
  All Data | 44.9 (26.0)
  0 Positive Nodes | 47.7 (29.0)
  1-3 Positive Nodes | 43.8 (23.8)
  3+ Positive Nodes | 42.6 (27.4)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); Kruskal-Wallis one-way ANOVA was used to test whether there was a difference in %SUVmax (FLT1-FLT2) among LN statuses. H0: no difference between the 3 LN status; Test type: Superiority or Other; p = 0.86, Kruskal-Wallis; two-sided p value from Kruskal-Wallis one-way ANOVA

9. Secondary Outcome: %Change SUVmax From FLT1-FLT3 to Predict Lymph Node Status at Surgery
Description: %change in SUVmax from FLT1-FLT3 will be compared by lymph node status at surgery For the purposes of reporting, %change in SUVmax from FLT1-FLT3 will be consider the outcome.
Time Frame: Baseline (FLT-1) and post-NAC (FLT-3)
Population: Data on 30 patients with FLT3 were available for histopathological LN evaluation after NAC: 11 with negative nodes, 13 with 1-3 LN metastases and 6 with >3 LN metastases
Measure: Mean (Standard Deviation); unit: percent change in SUVmax from FLT1-FLT3
Arm/Group | Diagnostic (18F-FLT)
Number analyzed (Participants) | 30
percent change in SUVmax from FLT1-FLT3
  All Data | 71.4 (29.1)
  0 Positive Nodes | 65.2 (42.2)
  1-3 Positive Nodes | 77.6 (18.1)
  3+ Positive Nodes | 69.5 (19.5)
Statistical Analysis 1: Comparison: Diagnostic (18F-FLT); Test type: Superiority or Other; p = 0.67, Kruskal-Wallis — two-sided p value from Kruskal-Wallis one-way ANOVA

ADVERSE EVENTS:
Arm/Group | Diagnostic (18F-FLT)
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 8/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (18F-FLT) (N=90)
Flushing (General disorders) | 2 (3)
Paresthesia (General disorders) | 2 (2)
Peripheral sensory neopathy (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Wound Infenction (General disorders) | 1 (1)
Nail discoloration (General disorders) | 1 (1)
Pain in extremity (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (Psychiatric disorders) | 1 (1)
Insomnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less